CLINICAL TRIAL: NCT03800550
Title: A Phase 1, Open-label, Randomized, Crossover Study to Assess the Drug-Drug Interaction Between Bedaquiline and Clarithromycin in Healthy Adult Volunteers
Brief Title: A Study to Assess the Drug-Drug Interaction Between Bedaquiline and Clarithromycin in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CR108570; 2018-004302-25 (EudraCT Number); TMC207NTM1001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2019-01-09; First posted 2019-01-11 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy
MeSH Terms: interventions — bedaquiline; Clarithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Sequence 1: Bedaquiline and Clarithromycin (Experimental): Participants will receive bedaquiline on Day 1 in Period 1, followed by clarithromycin on Days 1-14 and bedaquiline on Day 5 in Period 2. There will be washout period of at least 28 days starting on Day 1.
  Interventions: Drug: Bedaquiline; Drug: Clarithromycin
- Treatment Sequence 2: Clarithromycin and Bedaquiline (Experimental): Participants will receive clarithromycin on Days 1-14 and bedaquiline on Day 5 in Period 1, followed by bedaquiline on Day 1 in Period 2. There will be a washout period of at least 28 days starting after bedaquiline administration on Day 5.
  Interventions: Drug: Bedaquiline; Drug: Clarithromycin

INTERVENTIONS:
Drug: Bedaquiline — Bedaquiline tablet will be administered, orally.
Drug: Clarithromycin — Clarithromycin tablet will be administered, orally.

SUMMARY:
The purpose of this study is to assess the effect of steady-state clarithromycin once every 12 hour on the pharmacokinetic parameters of bedaquiline and its active metabolite M2 after a single dose of bedaquiline.

ELIGIBILITY:
Inclusion Criteria:

* A female participant must have a negative highly sensitive serum (beta-human chorionic gonadotropin [beta-hCG]) pregnancy test at screening and on Day -1 in each treatment period
* Contraceptive use by women should be consistent with local regulations regarding the use of contraceptive methods for participants participating in clinical studies
* A female participant must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for at least 90 days after receiving the last dose of bedaquiline
* During the study and for a minimum of at least 90 days after receiving the last dose of bedaquiline: a) A male participant must wear a condom when engaging in any activity that allows for passage of ejaculate to another person (male participants should also be advised of the benefit for a female partner to use a highly effective method of contraception as condom may break or leak. b) A male participant must agree not to donate sperm for the purpose of reproduction
* Body mass index (BMI between 18.0 and 30.0 kilogram (kg) per meter square (inclusive), and body weight not less than 50 kg at screening

Exclusion Criteria:

* Participant has history or current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), lipid abnormalities, significant pulmonary disease (including bronchospastic respiratory disease), diabetes mellitus, hepatic or renal insufficiency (for example, estimated creatinine clearance below 60 milliliter per minute [mL/min] at screening), gastrointestinal disease (such as significant diarrhea, gastric stasis, or constipation that in the investigator's opinion could influence drug absorption or bioavailability), thyroid disease, neurologic or psychiatric disease, infection, or any other illness that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* Participant with a past history of heart arrhythmias (extrasystoles or tachycardia at rest), or history of risk factors for Torsade de Pointes syndrome (for example, hypokalemia, or family history of long QT syndrome). Family history of sudden unexplained death (including sudden infant death syndrome in a first-degree relative (that is, sibling, offspring, or biological parent). Ongoing bradyarrhythmias or ongoing hypothyroidism (confirmed by elevated thyroid-stimulating hormone [TSH] level)
* Participant with any history of clinically significant skin disease such as, but not limited to, dermatitis, eczema, drug rash, psoriasis, food allergy, or urticaria
* Participant has taken any disallowed therapies before the planned first intake of study drug
* Participant has a history of drug or alcohol abuse according to Diagnostic and Statistical Manual of Mental Disorders (5th edition) criteria within 5 years before screening or positive test result(s) for alcohol and/or drugs of abuse (including barbiturates, opiates, cocaine, amphetamines, methadone, benzodiazepines, methamphetamine, tetrahydrocannabinol, phencyclidine, and tricyclic antidepressants) at screening and on Day 1 of each treatment period

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2019-02-13 (Actual); Primary Completion 2019-06-04 (Actual); Study Completion 2019-06-04 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Analyte Concentration (Cmax) of Bedaquiline and its Metabolite (M2) | Pre-dose, 1, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 120, 168, and 240 hours Post-dose
  Cmax is the maximum observed analyte concentration.
Minimum Observed Analyte Concentration (Cmin) of Bedaquiline and its Metabolite (M2) | Pre-dose, 1, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 120, 168, and 240 hours Post-dose
  Cmin is the minimum observed analyte concentration.
Area Under the Analyte Concentration versus Time Curve (AUC) From Time of Administration up to 72 Hours Post Dosing (AUC72h) of Bedaquiline and its Metabolite (M2) | Pre-dose, 1, 2, 3, 4, 5, 6, 8, 12, 24, 48, and 72 hours Post-dose
  AUC72h is the area under the analyte concentration versus time curve (AUC) from time of administration up to 72 hours post dosing, calculated by linear-linear trapezoidal summation.
Area Under the Analyte Concentration versus Time Curve (AUC) From Time of Administration up to 240 Hours Post Dosing (AUC240h) of Bedaquiline and its Metabolite (M2) | Pre-dose, 1, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 120, 168, and 240 hours Post-dose
  AUC240h is the area under the analyte concentration-time curve from time 0 to 240 hours, calculated by linear-linear trapezoidal summation.

SECONDARY OUTCOMES:
Cmax of Clarithromycin and its Metabolite 14-OH-Clarithromycin | Pre-dose, 1, 2, 3, 4, 5, 6, 8, and 12 hours Post-dose
  Cmax is the maximum observed analyte concentration.
Time to Reach Maximum Observed Analyte Concentration (Tmax) of Clarithromycin and its Metabolite 14-OH-Clarithromycin | Pre-dose, 1, 2, 3, 4, 5, 6, 8, and 12 hours Post-dose
  Tmax is the actual sampling time to reach the maximum observed analyte concentration.
Cmin of Clarithromycin and its Metabolite 14-OH-Clarithromycin | Pre-dose, 1, 2, 3, 4, 5, 6, 8, and 12 hours Post-dose
  Cmin is the minimum observed analyte concentration.
Area Under the Analyte Concentration versus Time Curve (AUC) From Time of Administration up to 12 Hours Post Dosing (AUC12h) of Clarithromycin and its Metabolite 14-OH-Clarithromycin | Pre-dose, 1, 2, 3, 4, 5, 6, 8, and 12 hours Post-dose
  AUC12h is the area under the analyte concentration versus time curve (AUC) from time of administration up to 12 hours post dosing, calculated by linear-linear trapezoidal summation.
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Up to 90 days
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- SGS Life Science Services, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency